CLINICAL TRIAL: NCT04447157
Title: The Efficacy of a 6-point Transscleral Suture Fixation of a 3-looped Haptics PC-IOL Implantation Through Scleral Pockets for Surgical Management for Microspherophakia
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: xuwen2020-465
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Microspherophakia
MeSH Terms: conditions — Microspherophakia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Microspherophakia: This is a non-interventional study(NIS). All the patients diagnosed as microspherophakia are included in the study and recieved intraocular lens implantation

SUMMARY:
By comparing the preoperative data and postoperative data of 9 patients of microspherophakia, we concluded that the 6-point transscleral suture fixation of a 3-looped haptics posterior chamber intraocular lens (PC-IOL) through scleral pockets was a feasible method of PC-IOL implantation in the surgical treatment of microspherophakia.

ELIGIBILITY:
Inclusion Criteria:

* Microspherophakia was diagnosed and lens diameter<9mm;
* The lens subluxation was beyond the range of one quadrant and glasses cannot correct the vision;
* Lens dislocated into the anterior chamber;
* Lens dislocation caused elevated intraocular pressure (IOP);
* The lens contacted the corneal endothelium;
* Cataract;
* Corneal endothelial cell density>1000/mm2;
* The fundus was normal without retinal detachment, severe macular disease and optic nerve atrophy；
* There was possible improvement in postoperative visual acuity measured by retinometer.

Exclusion Criteria:

* The lens is centered and the position of the lens is stable;
* Glasses can correct the vision obviously;
* The reason for the elevated IOP was independent with the lens;
* A high possibility of corneal decompensation after surgery;
* Fundus function was poor and it is not expected to improve the vision after surgery;
* Combined with other ocular diseases which were not suitable for IOL implantation;
* Combined with a systemic disease that the patient cannot tolerate the surgery.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A retrospective study was conducted on 9 patients (18 eyes) diagnosed with microspherophakia in Eye Center of the Second Affiliated Hospital, Zhejiang University School of Medicine from July 2016 to April 2020.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Visual function | 6 month postoperation
  Best corrected visual acuity (BCVA) measured using a decimal chart
Visual function | 6 month postoperation
  uncorrected distance visual acuity (UDVA) measured using a decimal chart
Intraocular pressure | 6 month postoperation
  intraocular pressure measured using non-contact tonometer
PCIOL tilt degree | 6 month postoperation
  PCIOL tilt degree measured using Ultrasound biomicroscope
PCIOL decentration distance | 6 month postoperation
  PCIOL decentration distance measured using Ultrasound biomicroscope
Endothelial cell density | 6 month postoperation
  Endothelial cell density was measured by specular microscopy
Anterior chamber depth | 6 month postoperation
  Anterior chamber depth measured using Ultrasound biomicroscope